CLINICAL TRIAL: NCT01289379
Title: The Effect of High Frequency Jet Ventilation (HFJV)on Pneumoperitoneum Induced Cardiovascular Changes, During Laparoscopic Surgery.
Brief Title: The Effect of High Frequency Jet Ventilation (HFJV)During Laparoscopic Operations
Acronym: HFJV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Other Study IDs: Bickel-HFJV
Record Dates: First submitted 2010-10-19; First posted 2011-02-03 (Estimated); Last update posted 2011-02-03 (Estimated); Status verified 2011-02

CONDITIONS: Cholecystolithiasis
Keywords: pneumoperitoneum; laparoscopy; HFJV; cardiovascular; Symptomatic
MeSH Terms: conditions — Cholecystolithiasis; Pneumoperitoneum | interventions — High-Frequency Jet Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HFJV (Experimental)
  Interventions: Procedure: High Frequency Jet Ventilation; Procedure: HFJV

INTERVENTIONS:
Procedure: High Frequency Jet Ventilation
Procedure: HFJV

SUMMARY:
Investigators conducted a randomised perspective study to determine whether the use of HFJV instead of conventional mechanical ventilation will reduce the adverse cardiovascular effects of pneumoperitoneum during laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients, undergoing laparoscopic surgery for Symptomatic cholecystolithiasis.

Exclusion Criteria:

* ASA 3 and 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Cardiac functionality (Cardiac output,VOLUME)
  Cardiac functionality (Cardiac output,VOLUME)

CONTACTS AND LOCATIONS:
Locations (1):
- Western Galilee Hospital, Nahariya, Israel